CLINICAL TRIAL: NCT05808439
Title: Endovascular Abdominal Aortic Aneurysm Repair
Brief Title: Endovascular Repair of AAA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Mohamed Awad Hassan, Assistant lecturer, Assiut University
Other Study IDs: Endovascular repair of AAa
Record Dates: First submitted 2023-03-30; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: On Abdominal Aortic Aneurysms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We study differen t endovascular techniques as an alternative to surgical reconstruction to repair AAAS regarding ; success rates, 30-day mortality, endoleak events secondary intervention rates

ELIGIBILITY:
Inclusion Criteria:

* Older than 18

Exclusion Criteria:

* inflammatory or mycotic AAA

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient older than 18 years
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-04-15 (Estimated); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
30 day mortality | 30 days
  Total death

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Assuit, Asyut, Assuit
  - Assuit, Asyut